CLINICAL TRIAL: NCT06105216
Title: The Effect of Crossword and Word Search Puzzles on Nursing Students' Parenteral Medication Administration Knowledge: A Randomized Controlled Study
Brief Title: The Effect of Crossword and Word Search Puzzles on Nursing Students' Parenteral Medication Administration Knowledge
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Evrim Eyikara (Other)
Responsible Party: Sponsor-Investigator, Evrim Eyikara, Director, Gazi University
Organization: Gazi University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2023-253
Record Dates: First submitted 2023-10-16; First posted 2023-10-27 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Nursing Education; Medicatioon Administration Knowledge; Puzzle

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental)
  Interventions: Other: Crossword and word search puzzles
- Control Group (No Intervention)

INTERVENTIONS:
Other: Crossword and word search puzzles — Students in the intervention group received hard copies of the puzzles at the end of the laboratory practice.
  Arms: Intervention Group

SUMMARY:
This study was conducted in a pretest-posttest parallel-group, randomized controlled design.The population of the study consisted of students (n=220) enrolled in the Fundamentals of Nursing course at the Faculty of Nursing of a public university in the 2022-2023 academic year.According to the exclusion criteria, 56 students were excluded from the study. One hundred sixty-four students who met the inclusion criteria were randomized to the intervention I (n = 82) and control groups (n = 82) by stratified block randomization after the completion of baseline measures. The study was completed with 164 students. The theoretical lecture was carried out by a researcher who was an expert faculty member in Fundamentals of Nursing. All students completed the pretest after attending the theoretical lecture. In the laboratory practice after the theoretical lecture, all students were divided into small groups and practiced parenteral medication administration skills one-to-one under the guidance of the instructor. Students in the intervention group received hard copies of the puzzles at the end of the laboratory practice. All students completed the posttest again at the end of the laboratory practice. Students were supervised during the tests and were not allowed to consult any books, the internet, or any other source of information.

ELIGIBILITY:
Inclusion Criteria:

(1) Register for the Fundamentals of Nursing course for the first time.

Exclusion Criteria:

1. not communicate in Turkish
2. graduate from any health-related university in the past.

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 220 (Actual)
Dates: Start 2023-04-26 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Medication Administration Knowledge Questionnaire | Through study completion, an average of 2 months
  Higher scores mean a better knowledge about parenteral medication administration (minimum score is 0, maximum score is 100)

CONTACTS AND LOCATIONS:
Locations (1):
- Gülcan Eyüboğlu, Ankara, Yenimahalle, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No